CLINICAL TRIAL: NCT04240743
Title: Comparison of Intramedullary and Extramedullary Fixation of Basicervical Fractures of the Femur in the Elderly: a Prospective, Randomized Controlled Trial
Brief Title: Fixation Methods of Basicervical Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Huseyin Bilgehan Cevik, Orthopaedic surgeon, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/514/74/7
Record Dates: First submitted 2020-01-17; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hip Fractures; Osteoporotic Fractures
Keywords: Basicervical; Cervicobasiler; Hip; Fracture; Prospective randomized
MeSH Terms: conditions — Hip Fractures; Osteoporotic Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cephalomedullary nail (Active Comparator): Cephalomedullary nails was inserted and fixed to the femoral head. In this study, all patients were treated with short nails (Profin®, TST).
  Interventions: Device: cephalomedullary nail; Device: sliding hip screw
- sliding hip screw (Active Comparator): Sliding hip screws was inserted and fixed to the femoral head. In this study, all patients were treated with a side plate with three holes (DHS plate, TST).
  Interventions: Device: cephalomedullary nail; Device: sliding hip screw

INTERVENTIONS:
Device: cephalomedullary nail — For patients in the cephalomedullary nail group, an incision was made in the gluteal area from the tip of the greater trochanter in proximal orientation. A guidewire was placed into the medullary canal from slightly medial to the exact tip of the greater trochanter. The entry point of the greater trochanter and proximal medullary canal were reamed. The cephalomedullary nail was then inserted and fixed to the femoral head with a double screw. The cephalomedullary nail was then locked distally using a guide arm. These cephalomedullary nails were not locked proximally to maintain dynamization and to allow compression across the basicervical fracture line.
Device: sliding hip screw — For patients in the sliding hip screw group, a lateral incision was made over the lateral proximal aspect of the femur. Under fluoroscopic guidance, the lag screw was placed centrally in the femoral head over the guidewire. A side plate with three holes was then attached to the hip screw.

SUMMARY:
This prospective, randomized study included patients aged over 65 years with basicervical fracture of femur from January 2016 to January 2018. The permuted block randomization method was used to randomize participants into groups. The patients were allocated to one of two groups treated via cephalomedullary nail (CMN) or sliding hip screw (SHS). Functional and radiological evaluations was included the mobility score, Harris hip score, modified Barthel index, the Singh index, the tip-apex distance, and fracture settling.

DETAILED DESCRIPTION:
Approval for this prospective randomized study was granted by the Local Ethics Review Board and all procedures were performed in accordance with the ethical standards of the Declaration of Helsinki (1964). Patients with a basicervical femur fracture were identified on admission to the Emergency Department of our tertiary hospital from January 2016 to January 2018. Patients with scheduled surgery who met the inclusion criteria and provided written informed consent were included in the study.

Patients were randomly allocated to a study group by permuted blocks of randomly mixed sizes and stratification according to the type of surgery (CMN or SHS). Randomization was applied using pre-prepared randomization cards, which were placed in opaque sealed envelopes and given to the surgeons to open just prior to surgery, and the designated procedure was then performed.

ELIGIBILITY:
Inclusion Criteria:

* basicervical fracture,
* age of ≥65 year,
* an isolated fracture,
* the ability to walk independently (with or without an aid) prior to fracture,
* a fracture that had occurred less than one week prior to admission.

Exclusion Criteria:

* history of ipsilateral femoral fracture,
* a fracture due to malignancy,
* limited life expectancy due to medical comorbidities,
* any contraindication to surgery,
* diagnosed dementia,
* any other traumatic fracture on admission.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
mobility score | 12 months
  Functional outcome was assessed by the mobility score of Parker and Palmer (Parker MJ, Palmer CR (1993) A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br 75: 797-798), which uses a nine-point scale.
Harris hip score | 12 months
  Hip function was rated with Harris Hip Score. The score has a maximum of 100 points (best possible function), covering pain (1 item, 0-44 points), function and activities (7 items, 0-47 points), and range of motion and absence of deformity (3 items, 0-9 points).
modified Barthel index | 12 months
  Barthel Index (Mahoney FI, Barthel DW (1965) Functional evaluation: the Barthel Index. A simple index of independence useful in scoring improvement in the rehabilitation of the chronically ill. Md State Med J 13:61-65), which measures the level of functional independence for 10 activities of daily living and ranges from 0 to 100.
the tip-apex distance | 12 months
  It uses a numerical value (the distance between tip of screw and subchondral area) to show placement of the screw in the head: higher values indicating higher likelihood of fixation failure by extrusion of the screw.
fracture settling | 12 months
  It uses a numerical value to show placement of shortening of the fractured femoral neck in time

IPD SHARING:
Plan to Share IPD: Undecided